CLINICAL TRIAL: NCT04726787
Title: RadiothErapy priMIng for CAR-T
Acronym: REMIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/137861
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bridging Radiotherapy (Experimental): Disease areas requiring effective long-term control will receive full-dose radiotherapy (20-30Gy/5-15#); other areas will receive low dose (4Gy/2#)
  Interventions: Radiation: Bridging Radiotherapy

INTERVENTIONS:
Radiation: Bridging Radiotherapy — Bridging Radiotherapy will start immediately after leukapheresis and before Tisagenlecleucel treatment

SUMMARY:
The REMIT trial will investigate radiotherapy as a preferred bridging method prior to Tisagenlecleucel infusion in patients with relapsed or refractory Diffuse Large B Cell Lymphoma

DETAILED DESCRIPTION:
The REMIT Trial is an open label, single arm phase IIa study investigating Radiotherapy as preferred bridging method prior to Tisagenlecleucel treatment in patients with relapsed or refractory Diffuse Large B Cell Lymphoma approved to receive CD19 CAR-T cells as per their licensed indication.

The trial will recruit 20 patients who have been approved to receive Tisagenlecleucel treatment and where the tumour is amendable to radiotherapy as per standard of care.

Trial subjects (patients) during a 14 day screening phase will have their metabolic tumour burden assessed by PET-CT and bridging radiotherapy will be planned. Bridging radiotherapy will commence immediately after leukapheresis with dose adjustments according to disease burden and localisation.

Disease areas requiring effective long-term control will receive full dose radiotherapy, 20 - 30Gy /5-15# and other areas will receive low dose radiotherapy, 4Gy / 2# for optimal tumour debulking and priming effects.

Standard lymphodepletion will be given day -5 to day -3 followed by Tisagenlecleucel infusion on day 0. A window of 14-21 days will be left from last dose of radiotherapy and day 0.

Patients will be followed up at 3 and 6 months after Tisagenlecleucel infusion for a minimum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥ 18 years
3. Histologically proven DLBCL, including transformed follicular or marginal zone lymphoma
4. Measurable disease on cross-sectional imaging that is at least 1.5cm in the longest diameter and measurable in two perpendicular dimensions
5. Relapsed/refractory after 2 or more standard immuno-chemotherapies
6. Approved to receive Tisagenlecleucel as per the licenced indication
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Disease accessible for repeat biopsies (Selected patients only)
9. Disease amenable to radiotherapy as assessed by the treating clinical oncologist
10. Willing and able to comply with the requirements of the protocol, including contraceptive advice as per the protocol

Exclusion Criteria:

1. Prior radiotherapy at location/dose that would interfere with application of radiotherapy or outcome measures in this trial
2. Women who are pregnant or breast feeding
3. Previous therapy with any genetically modified autologous or allogeneic T-cell immunotherapy, unless treated with doses of genetically modified autologous or allogeneic T-cell immunotherapy within an abandoned dosing cohort in a first in human dose-escalation phase I clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients starting lymphodepletion on the planned start date without delay | From planned start date of lymphodepletion until actual start date of lymphodepletion, assessed up to 2 weeks
  To evaluate whether there is any delay in patients starting lymphodepletion

SECONDARY OUTCOMES:
Best overall response after Tisagenlecleucel infusion as per International Working Group 2014 criteria | After Tisagenlecleucel infusion through to study completion, an average of 24 months
  Proportion of patients achieving a Complete Response (CR) or Partial Response (PR)
Overall response rate at 3 months and 6 months after Tisagenlecleucel infusion | At 3 and 6 months after Tisagenlecleucel infusion
  Overall response rate after Tisagenlecleucel infusion
Complete metabolic response at 3 months and 6 months after Tisagenlecleucel infusion | At 3 and 6 months after Tisagenlecleucel infusion
  Complete metabolic response after Tisagenlecleucel infusion
Duration of response | From initial response until the date of first documented disease progression, assessed up to 24 months
  Time from date of first response confirmation to the first date of progressive disease confirmation
Median progression free survival and progression free survival at 12 months | 12 months after Tisagenlecleucel infusion
  Progression Free Survival after Tisagenlecleucel infusion
Median event-free survival and event-free survival at 12 months | 12 months after Tisagenlecleucel infusion
  Event-free survival after Tisagenlecleucel infusion
Median overall survival and overall survival at 12 months | 12 months after Tisagenlecleucel infusion
  Overall Survival after Tisagenlecleucel infusion
Treatment emergent adverse events | From start of Tisagenlecleucel infusion until 30 days post Tisagenlecleucel infusion
  Adverse events being reported during and after treatment
Incidence of grade 3 or higher cytokine release syndrome and immune effector cell associated neurotoxicity syndrome | From start of Tisagenlecleucel infusion through to study completion, an average of 24 months
  Percentage of grade 3 or higher cytokine relapse syndrome and immune effector cell associated neurotoxicity syndrome events
Neutrophil levels at 1, 3, 6 months after Tisagenlecleucel infusion | At 1, 3 and 6 months after Tisagenlecleucel infusion
  Neutrophil counts to be reported after Tisagenlecleucel infusion
Platelet levels at 1, 3, 6 months after Tisagenlecleucel infusion | At 1, 3 and 6 months after Tisagenlecleucel infusion
  Platelet counts to be reported after Tisagenlecleucel infusion

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kuhnl, Study Chair — King's College Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - St James's University Hospital, Leeds
  - Kings College Hospital, London
  - Freeman Hospital, Newcastle